CLINICAL TRIAL: NCT01490294
Title: Multicenter, Double Blind, Randomized Dose Finding Study in Myocardial Perfusion MRI With Gadavist®1.0
Brief Title: Myocardial Perfusion MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 91054; 305501 (Other: Bayer Healthcare AG); 2005-005158-32 (EudraCT Number)
Record Dates: First submitted 2011-07-28; First posted 2011-12-12 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Myocardial Perfusion Imaging; Magnetic Resonance Imaging
Keywords: Cardiac MRI; gadobutrol
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) (Experimental): Participants received 1 i.v. bolus injections of Gadobutrol 0.01 mmol/kg body weight (BW) (0.01mL/kg) for stress magnetic resonance imaging (MRI) via a power injector at a rate of 3 mL/s. The second i.v. bolus injection of Gadobutrol 0.01 mmol/kg BW was given after a 10-15 minutes wash-out period of the stressor for the rest MRI.
  Interventions: Drug: Gadobutrol (Gadavist,Gadovist, BAY86-4875)
- Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) (Experimental): Participants received 1 i.v. bolus injections of Gadobutrol 0.025 mmol/kg BW (0.01mL/kg) for stress MRI via a power injector at a rate of 3 mL/s. The second i.v. bolus injection of Gadobutrol 0.025 mmol/kg BW was given after a 10-15 minutes wash-out period of the stressor for the rest MRI.
  Interventions: Drug: Gadobutrol (Gadavist,Gadovist, BAY86-4875)
- Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) (Experimental): Participants received 1 i.v. bolus injections of Gadobutrol 0.05 mmol/kg BW (0.01mL/kg) for stress MRI via a power injector at a rate of 3 mL/s. The second i.v. bolus injection of Gadobutrol 0.05 mmol/kg BW was given after a 10-15 minutes wash-out period of the stressor for the rest MRI.
  Interventions: Drug: Gadobutrol (Gadavist,Gadovist, BAY86-4875)
- Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) (Experimental): Participants received 1 i.v. bolus injections of Gadobutrol 0.1 mmol/kg BW (0.01mL/kg) for stress MRI via a power injector at a rate of 3 mL/s. The second i.v. bolus injection of Gadobutrol 0.1 mmol/kg BW was given after a 10-15 minutes wash-out period of the stressor for the rest MRI.
  Interventions: Drug: Gadobutrol (Gadavist,Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist,Gadovist, BAY86-4875) — 0.01 mmol/kg BW (0.01 mL/kg) for stress MRI and 0.01 mmol/kg BW (0.01 mL/kg) for rest MRI (total dose 0.02 mmol/kg)
  Arms: Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875)
Drug: Gadobutrol (Gadavist,Gadovist, BAY86-4875) — 0.025 mmol/kg BW (0.025 mL/kg) for stress MRI and 0.025 mmol/kg BW (0.025 mL/kg) for rest MRI (total dose 0.05 mmol/kg)
  Arms: Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875)
Drug: Gadobutrol (Gadavist,Gadovist, BAY86-4875) — 0.05 mmol/kg BW (0.05 mL/kg) for stress MRI and 0.05 mmol/kg BW (0.05 mL/kg) for rest MRI (total dose 0.1 mmol/kg)
  Arms: Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875)
Drug: Gadobutrol (Gadavist,Gadovist, BAY86-4875) — 0.1 mmol/kg BW (0.1 mL/kg) for stress MRI and 0.1 mmol/kg BW (0.1 mL/kg) for rest MRI (total dose 0.2 mmol/kg)
  Arms: Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)

SUMMARY:
The object of this study is to compare four different dosages of Gadavist 1.0 in cardiac Magnetic Resonance Tomography (MRT) imaging with the imaging results of a cardiac SPECT examination in terms of diagnostic quality.

For this purpose Gadavist dosages of 0.01 mmol/kg, 0.025 mmol/kg, 0.05 mmol/kg or 0.1mmol/kg body weight are administered. A study participant receives the respective dose twice i.e. at rest and at stress using Adenosine (which puts circulation into a state of stress similar to that of physical exercise). The time between both injections is 10-15 min.

The total imaging time is about 45 min.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any ethnic group with reversible focal hypoperfusion in at least 2 adjoining segments in SPECT
* The SPECT examination had been performed within 4 weeks prior to the MRI examination and had been performed for clinical reasons only

Exclusion Criteria:

* Generalized myocardial hypoperfusion (e.g. severe 3 vessel disease)
* Recent myocardial infarction (MI) (within 1 week prior to the study procedure)
* Event that significantly altered cardiac performance between SPECT and MRI imaging, e.g. myocardial infarction, unstable angina, alteration of cardiac medication
* Non-sinus rhythm
* Sinus node disease or symptomatic bradycardia
* Second or third degree atrial ventricular (AV) block
* Complete left bundle branch block (LBBB)
* Known congenital long QT syndrome or a family history of congenital long QT syndrome
* Known previous arrhythmias on drugs that prolong cardiac repolarization
* Uncorrected hypokalemia
* Uncontrolled hypertension (e.g. systolic blood pressure >185 mm Hg, diastolic blood pressure >110 mm Hg)
* Baseline hypotension (e.g. mean arterial pressure <60 mm Hg)
* Ejection fraction below 35%
* Cardiomyopathy, congenital heart defect or higher degree valvular pathology
* Coronary artery stent placement within 4 weeks prior to the MRI procedure
* Previous heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2004-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Pölten, Austria
- Germany (9):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Bad Oeynhausen, North Rhine-Westphalia
  - Bonn, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Berlin
- Krakow, Poland
- Switzerland (2):
  - Basel, Canton of Basel-City
  - Lugano, Canton Ticino

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Started | 58 | 60 | 59 | 55
Participant Received Treatment | 54 | 60 | 58 | 54
Completed | 53 | 60 | 58 | 54
Not Completed | 5 | 0 | 1 | 1
Not completed — Prematurely discontinuation | 4 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) | Total
Number analyzed (Participants) | 54 | 60 | 58 | 54 | 226
Age, Continuous [Median (Full Range); unit: Years] — The study was planned and conducted to provide data for 4 different increasing doses of Gadobutrol. Therefore, the age was not calculated over all four dose groups of Gadobutrol.
  Years | 62.0 [29 to 78] | 61.5 [32 to 83] | 64.5 [39 to 81] | 61.0 [35 to 79] | 62.0 [29 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 17 | 19 | 70
  Male | 39 | 41 | 41 | 35 | 156
History of myocardial infarction [Number; unit: Participants]
  No | 34 | 42 | 43 | 37 | 156
  Yes | 20 | 17 | 15 | 15 | 67
  Unknown | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Agreement Between Gadobutrol Perfusion Magnetic Resonance Imaging (MRI) (Blinded Reading) and SPECT (Central Reading) Regarding the Diagnosis for Detection of Cardiac Perfusion Deficits Based on Myocardial Regions
Description: Rest and stress perfusion Magnetic Resonance (MR) images were evaluated by 3 independent blinded readers for presence/absence of cardiac perfusion deficits in 3 myocardial regions representing the 3 coronary territories/arteries (left anterior decendent [LAD], left circumflex [LCX], right coronary artery [RCA]). Data were compared to the corresponding regional data from Single Photon Emission Computer Tomography (SPECT). The number of regional assessments was calculated by multiplication of the number of participants with the number of the blinded readers and number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: Per protocol set (PPS)
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional assessments
Groups:
- Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875): Participants received 1 i.v. bolus injections of Gadobutrol 0.01 mmol/kg BW (0.01mL/kg) for stress MRI via a power injector at a rate of 3 mL/s. The second i.v. bolus injection of Gadobutrol 0.01 mmol/kg BW was given after a 10-15 minutes wash-out period of the stressor for the rest MRI.
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Regional assessments) | 396 | 513 | 477 | 477
Percent regional assessments
  Disagreement | 58.8 | 44.1 | 36.7 | 40.3
  Agreement | 41.2 | 55.9 | 63.3 | 59.7

2. Primary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading) and SPECT (Central Reading) Regarding the Diagnosis for Detection of Cardiac Perfusion Deficits Based on Myocardial Segments
Description: Rest and stress perfusion MR images were evaluated by 3 independent blinded readers for presence/absence of cardiac perfusion deficits in 16 myocardial segments (defined according to the American Heart Association). These data were compared to the corresponding segmental data from SPECT. The number of segmental assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: Per protocol set (PPS)
Measure: Number; unit: Percent segmental assessment
Units Other Than Participants: Segmental Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segmental Assessment) | 2112 | 2736 | 2544 | 2544
Percent segmental assessment
  Disagreement | 51.1 | 39.4 | 34.5 | 34.1
  Agreement | 48.9 | 60.6 | 65.5 | 65.9

3. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Clinical Evaluation) and SPECT (Central Reading) Regarding the Diagnosis for Detection of Cardiac Perfusion Deficits Based on Myocardial Regions
Description: Rest and stress perfusion MR images were evaluated by the respective clinical investigator for presence/absence of cardiac perfusion deficits in 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). These data were compared to the corresponding regional data from SPECT. The number of regional assessments was calculated by multiplication of the number of participants with the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Regional Assessments) | 132 | 171 | 153 | 153
Percent regional assessments
  Disagreement | 48.5 | 39.2 | 35.2 | 37.7
  Agreement | 51.5 | 60.8 | 64.8 | 62.3

4. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Clinical Evaluation) and SPECT (Central Reading) Regarding the Diagnosis for Detection of Cardiac Perfusion Deficits Based on Myocardial Segments
Description: Rest and stress perfusion MR images were evaluated by the respective investigator for presence/absence of cardiac perfusion deficits in 16 myocardial segments (defined according to the American Heart Association). These data were compared to the corresponding segmental data from SPECT. The number of segmental assessments was calculated by multiplication of the number of participants with the number of the myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segmental Assessments) | 704 | 912 | 848 | 848
Percent segmental assessments
  Disagreement | 39.3 | 30.4 | 28.7 | 33.3
  Agreement | 60.7 | 69.6 | 71.3 | 66.7

5. Secondary Outcome: Diagnosis 'Scar': Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading) and SPECT (Central Reading) Regarding the Diagnosis Scar Based on Myocardial Regions
Description: Rest and stress perfusion MR images were evaluated by 3 independent blinded readers for presence/absence and characterization of cardiac perfusion deficits as "scar" in the 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). These data were compared to the corresponding regional SPECT diagnosis of 'scar'. The number of regional assessments is defined as the number of regions with diagnosis 'scar' assessed by at least 1 blinded reader.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. Only patients with the finding "scar" in at least 1 region in SPECT were included.
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 12 | 19 | 13 | 19
Number analyzed (Regional Assessments) | 48 | 72 | 42 | 96
Percent regional assessments
  Disagreement | 81.3 | 80.6 | 83.3 | 86.5
  Agreement | 18.8 | 19.4 | 16.7 | 13.5

6. Secondary Outcome: Diagnosis "Scar": Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading) and SPECT (Central Reading) Regarding the Diagnosis "Scar" Based on Myocardial Segments
Description: Rest and stress perfusion MR images were evaluated by 3 independent blinded readers for presence/absence and characterization of cardiac perfusion deficits as "scar" in 16 myocardial segments (defined according to the American Heart Association). These data were compared to corresponding segmental SPECT diagnosis of "scar". The number of segmental assessments is defined as the number of segments with diagnosis "scar" assessed by at least 1 blinded reader.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. Only patients with the finding "scar" in at least 1 segment in SPECT were included.
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 12 | 19 | 13 | 19
Number analyzed (Segmental Assessments) | 129 | 147 | 111 | 195
Percent segmental assessments
  Disagreement | 88.4 | 85.7 | 82.0 | 90.8
  Agreement | 11.6 | 14.3 | 18.0 | 9.2

7. Secondary Outcome: Diagnosis "Scar": Percentage Agreement Between Gadobutrol Perfusion MRI (Clinical Evaluation) and SPECT (Central Reading) Regarding the Diagnosis "Scar" Based on Myocardial Regions
Description: Rest and stress perfusion MR images were evaluated by the respective clinical investigator for presence/absence and characterization of cardiac perfusion deficits as "scar" in the 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). These data were compared to the corresponding regional SPECT diagnosis of "scar". The number of regional assessments is defined as the number of segments with diagnosis "scar" assessed by the investigator.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: as for outcome 5
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 9 | 18 | 13 | 16
Number analyzed (Regional Assessments) | 11 | 25 | 17 | 21
Percent regional assessments
  Disagreement | 81.8 | 76.0 | 76.5 | 85.7
  Agreement | 18.2 | 24.0 | 23.5 | 14.3

8. Secondary Outcome: Diagnosis "Scar": Percentage Agreement Between Gadobutrol Perfusion MRI (Clinical Evaluation) and SPECT (Central Reading) Regarding the Diagnosis "Scar" Based on Myocardial Segments
Description: Rest and stress perfusion MR images were evaluated by the respective clinical investigator for presence/absence and characterization of cardiac perfusion deficits as "scar" in 16 myocardial segments (defined according to the American Heart Association). These data were compared to the corresponding segmental SPECT diagnosis of "scar". The number of segmental assessments is defined as the number of segments with diagnosis "scar" assessed by the investigator.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: as for outcome 6
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 9 | 18 | 13 | 16
Number analyzed (Segmental Assessments) | 22 | 46 | 33 | 50
Percent segmental assessments
  Disagreement | 86.4 | 84.8 | 69.7 | 88.0
  Agreement | 13.6 | 15.2 | 30.3 | 12.0

9. Secondary Outcome: Diagnosis "Ischemia": Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading) and SPECT (Central Reading) Regarding the Diagnosis of Ischemia Based on Myocardial Regions
Description: Rest and stress perfusion MR images were evaluated by 3 independent blinded readers for presence/absence and characterization of cardiac perfusion deficits as "ischemia" in the 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). These data were compared to the corresponding regional SPECT diagnosis of "ischemia".The number of regional assessments is defined as the number of regions with diagnosis "ischemia" assessed by at least 1 blinded reader.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. Only patients with the finding "ischemia" in at least 1 region in SPECT were included.
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 35 | 46 | 48 | 38
Number analyzed (Regional Assessments) | 198 | 228 | 216 | 213
Percent regional assessments
  Disagreement | 87.9 | 69.3 | 64.4 | 60.6
  Agreement | 12.1 | 30.7 | 35.6 | 39.4

10. Secondary Outcome: Diagnosis "Ischemia": Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading) and SPECT (Central Reading) Regarding the Diagnosis of Ischemia Based on Myocardial Segments
Description: Rest and stress perfusion MR images were evaluated by 3 independent blinded readers for presence/absence and characterization of cardiac perfusion deficits as "ischemia" in 16 myocardial segments (defined according to the American Heart Association). These data were compared to corresponding segmental SPECT diagnosis of "ischemia". The number of segmental assessments is defined as the number of segments with diagnosis "ischemia" assessed by at least 1 blinded reader.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. Only patients with the finding "ischemia" in at least 1 segment in SPECT were included.
Measure: Number; unit: Percent segmental assessment
Units Other Than Participants: Segmental Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 35 | 46 | 48 | 38
Number analyzed (Segmental Assessment) | 513 | 561 | 567 | 588
Percent segmental assessment
  Disagreement | 91.8 | 77.5 | 74.3 | 68.9
  Agreement | 8.2 | 22.5 | 25.7 | 31.1

11. Secondary Outcome: Diagnosis "Ischemia": Percentage Agreement Between Gadobutrol Perfusion MRI (Clinical Evaluation) and SPECT (Central Reading) Regarding the Diagnosis of Ischemia Based on Myocardial Regions
Description: Rest and stress perfusion MR images were evaluated by the respective clinical investigator for presence/absence and characterization of cardiac perfusion deficits as "ischemia" in the 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). These data were compared to the corresponding regional SPECT diagnosis of "ischemia". The number of regional assessments is defined as the number of regions with diagnosis "ischemia" assessed by the investigator.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: as for outcome 9
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 43 | 56 | 53 | 53
Number analyzed (Regional Assessments) | 74 | 96 | 89 | 90
Percent regional assessments
  Disagreement | 63.5 | 61.5 | 48.3 | 46.7
  Agreement | 36.5 | 38.5 | 51.7 | 53.3

12. Secondary Outcome: Diagnosis "Ischemia": Percentage Agreement Between Gadobutrol Perfusion MRI (Clinical Evaluation) and SPECT (Central Reading) Regarding the Diagnosis of Ischemia Based on Myocardial Segments
Description: Rest and stress perfusion MR images were evaluated by the respective clinical investigator for presence/absence and characterization of cardiac perfusion deficits as "ischemia" in 16 myocardial segments (defined according to the American Heart Association). These data were compared to corresponding segmental SPECT diagnosis of "ischemia". The number of segmental assessments is defined as the number of segments with diagnosis "ischemia" assessed by the investigator.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: as for outcome 10
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 43 | 56 | 53 | 53
Number analyzed (Segmental Assessments) | 186 | 222 | 221 | 232
Percent segmental assessments
  Disagreement | 77.4 | 66.7 | 58.4 | 58.2
  Agreement | 22.6 | 33.3 | 41.6 | 41.8

13. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading) and SPECT (Central Reading) Regarding a Detailed Diagnosis of Cardiac Perfusion Deficits i.e. Scar, Ischemia or a Mixture of Both, Based on Myocardial Regions
Description: Rest and stress perfusion MR images were evaluated by 3 independent blinded readers for detailed characterization of cardiac perfusion deficits i.e. scar, ischemia or mixture of both in 3 myocardial regions representing 3 coronary territories/arteries (LAD, LCX, RCA). MR data were compared to the corresponding regional data from SPECT. The number of regional assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Regional Assessments) | 396 | 513 | 477 | 477
Percent regional assessments
  Disagreement | 67.4 | 57.3 | 46.8 | 53.0
  Agreement | 32.6 | 42.7 | 53.2 | 47.0

14. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading) and SPECT (Central Reading) Regarding a Detailed Diagnosis of Cardiac Perfusion Deficits i.e. Scar, Ischemia or a Mixture of Both Based on Myocardial Segments
Description: Rest and stress perfusion MR images were evaluated by 3 independent blinded readers for detailed characterization of cardiac perfusion deficits i.e. scar, ischemia or mixture of both in 16 myocardial segments (defined according to the American Heart Association). MR data were compared to the corresponding segmental data from SPECT. The number of segmental assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent segmental assessment
Units Other Than Participants: Segmental Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segmental Assessment) | 2112 | 2736 | 2544 | 2544
Percent segmental assessment
  Disagreement | 53.8 | 42.7 | 36.8 | 37.3
  Agreement | 46.2 | 57.3 | 63.2 | 62.7

15. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Clinical Evaluation) and SPECT (Central Reading) Regarding a Detailed Diagnosis of Cardiac Perfusion Deficits i.e. Scar, Ischemia or a Mixture of Both Based on Myocardial Regions
Description: Rest and stress perfusion MR images were evaluated by the respective clinical investigator for detailed characterization of cardiac perfusion deficits i.e. scar, ischemia or mixture of both in 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). MR data were compared to the corresponding regional data from SPECT. The number of regional assessments was calculated by multiplication of the number of participants with the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Regional Assessments) | 132 | 171 | 159 | 159
Percent regional assessments
  Disagreement | 52.3 | 49.1 | 42.1 | 46.5
  Agreement | 47.7 | 50.9 | 57.9 | 53.5

16. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Clinical Evaluation) and SPECT (Central Reading) Regarding a Detailed Diagnosis of Cardiac Perfusion Deficits i.e. Scar, Ischemia or a Mixture of Both Based on Myocardial Segments
Description: Rest and stress perfusion MR images were evaluated by the respective clinical investigator for detailed characterization of cardiac perfusion deficits i.e. scar, ischemia or a mixture of both in 16 myocardial segments (defined according to the American Heart Association).MR data were compared to the corresponding segmental data from SPECT. The number of segmental assessments was calculated by multiplication of the number of participants with the number of the myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segmental Assessments) | 704 | 912 | 848 | 848
Percent segmental assessments
  Disagreement | 40.9 | 33.0 | 31.1 | 35.6
  Agreement | 59.1 | 67.0 | 68.9 | 64.4

17. Secondary Outcome: Percent Agreement Between Combined Gadobutrol Perfusion MRI (Perfusion Imaging and Delayed (DE) Imaging; Blinded Reading) and SPECT (Central Reading) Regarding a Detailed Diagnosis of Perfusion Deficits Based on Myocardial Regions
Description: Rest and stress perfusion and DE MR images were evaluated by 3 independent blinded readers regarding the detailed characterization of cardiac perfusion deficits i.e scar, ischemia or a mixture of both, in 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). MR data were compared to the corresponding regional data from SPECT. The number of regional assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Regional Assessments) | 396 | 513 | 477 | 477
Percent regional assessments
  Disagreement | 66.2 | 53.8 | 51.4 | 53.5
  Agreement | 33.8 | 46.2 | 48.6 | 46.5

18. Secondary Outcome: Percent Agreement Between Combined Gadobutrol Perfusion MRI (Perfusion Imaging and Delayed (DE) Imaging; Blinded Reading) and SPECT (Central Reading) Regarding a Detailed Diagnosis of Perfusion Deficits Based on Myocardial Segments
Description: Rest and stress perfusion and DE MR images were evaluated by 3 independent blinded readers regarding the detailed characterization of cardiac perfusion deficits i.e scar, ischemia or a mixture of both in 16 myocardial segments (defined according to the American Heart Association). MR data were compared to the corresponding segmental data derived from SPECT. The number of segmental assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segmental Assessments) | 2112 | 2736 | 2544 | 2544
Percent segmental assessments
  Disagreement | 48.5 | 41.2 | 35.6 | 35.3
  Agreement | 51.5 | 58.8 | 64.4 | 64.7

19. Secondary Outcome: Percentage of Artifacts in Gadobutrol Perfusion MRI (Blinded Reading) Based on Myocardial Segments
Description: Rest and stress MR images were evaluated by 3 independent blinded readers regarding the presence/absence of artifacts in 16 myocardial segments (according to the American Heart Association). The number of segmental assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percentage of segments with artifacts
Units Other Than Participants: Segments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segments) | 2112 | 2736 | 2544 | 2544
Percentage of segments with artifacts
  Missing | 1.8 | 1.4 | 2.8 | 1.5
  No | 66.3 | 62.7 | 62.1 | 66.3
  Yes | 31.9 | 35.9 | 35.0 | 32.2

20. Secondary Outcome: Percentage of Artifacts in Gadobutrol Perfusion MRI (Clinical Evaluation) Based on Myocardial Segments
Description: Rest and stress MR images were evaluated by the investigator regarding the presence/absence of artifacts in 16 myocardial segments (defined according to the American Heart Association). The number of segments with artifacts was calculated by multiplication of the number of participants with the number of the myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percentage of segments with artifacts
Units Other Than Participants: Segments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segments) | 704 | 912 | 848 | 848
Percentage of segments with artifacts
  No | 85.5 | 85.3 | 81.5 | 83.5
  Yes | 14.5 | 14.7 | 17.1 | 15.8
  Not assessable | 0.0 | 0.0 | 1.4 | 0.0
  Not determined | 0.0 | 0.0 | 0.0 | 0.7

21. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading, Based on Myocardial Regions) and Coronary Angiography (Central Reading) Regarding Detection of Significant Stenoses
Description: Rest and stress perfusion MR images were evaluated by 3 independent blinded readers for presence/absence of perfusion deficits in 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). These data were compared to coronary angiography regarding presence/absence of significant coronary artery stenosis of > 70%. The number of regional assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 18 | 30 | 25 | 34
Number analyzed (Regional Assessments) | 162 | 258 | 219 | 291
Percent regional assessments
  Disagreement | 50.6 | 48.1 | 38.8 | 32.3
  Agreement | 49.4 | 51.9 | 61.2 | 67.7

22. Secondary Outcome: Percentage Agreement Between the Semiquantitative Gadobutrol Perfusion MRI Parameter "Myocardial Perfusion Reserve Index (MPRI) " (Expert Evaluation) and Detection of Significant Stenoses by Coronary Angiography (MR Based on Myocardial Regions)
Description: MPRI was calculated for the upslope of the signal intensity /time curve on stress and rest perfusion MR images by an independent MR expert for 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). The upslope-value at post-stress was divided by the value at rest. MPRI <=1.5 (perfusion defect) and >1.5 (normal) were compared to coronary angiography regarding presence/absence of significant coronary artery stenosis of >70%. The number of regional assessments was calculated by multiplication of the number of participants with the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 18 | 30 | 25 | 34
Number analyzed (Regional Assessments) | 54 | 86 | 73 | 97
Percent regional assessments
  Disagreement | 53.7 | 40.7 | 60.3 | 56.7
  Agreement | 46.3 | 59.3 | 39.7 | 43.3

23. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI (Blinded Reading) and the Truth Panel Diagnosis (SoT) Regarding Perfusion Defects Based on Regions
Description: For patients undergoing coronary angiography additionally to SPECT, a Truth Panel with 2 cardiology experts was employed as SoT to come to a consensus diagnosis. Rest and stress MR images were evaluated by 3 independent blinded readers for presence/absence of perfusion defects in 3 myocardial regions representing the 3 arterial territories/arteries of the heart. These data were compared to the SoT diagnosis. The number of regional assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 23 | 35 | 29 | 36
Number analyzed (Regional Assessments) | 207 | 315 | 261 | 324
Percent regional assessments
  Disagreement | 62.8 | 51.4 | 53.6 | 40.7
  Agreement | 37.2 | 48.6 | 46.4 | 59.3

24. Secondary Outcome: Percentage Agreement Between the Semiquantitative Gadobutrol Perfusion MRI Parameter "Myocardial Perfusion Reserve Index (MPRI)" (Expert Evaluation) and SPECT (Central Reading) Based on Myocardial Regions
Description: MPRI was calculated as decribed in outcome measure 22 on stress and rest perfusion MR images by an independent MR expert for 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). MPRIs <= 1.5 (perfusion defect) and >1.5 (normal) were compared to presence/absence of perfusion defects in the regional data analysis from SPECT. The number of regional assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Regional Assessments) | 132 | 171 | 159 | 159
Percent regional assessments
  Disagreement | 62.1 | 60.8 | 59.1 | 66.0
  Agreement | 37.9 | 39.2 | 40.9 | 34.0

25. Secondary Outcome: Percentage Agreement Between the Semiquantitative Gadobutrol Perfusion MRI Parameter "Myocardial Perfusion Reserve Index (MPRI)" (Expert Evaluation) and SPECT (Central Reading) Based on Myocardial Segments
Description: MPRI was calculated as decribed in outcome measure 22 on stress and rest perfusion MR images by an independent MR expert for 16 myocardial segments (defined according to the American Heart Association). MPRIs <= 1.5 (perfusion defect) and >1.5 (normal) were then compared to presence/absence of perfusion defects in the segmental data from SPECT. The number of segmental assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segmental Assessments) | 704 | 912 | 848 | 848
Percent segmental assessments
  Disagreement | 69.6 | 57.0 | 48.9 | 49.4
  Agreement | 30.4 | 43.0 | 51.1 | 50.6

26. Secondary Outcome: Percentage Agreement Between the Visual (Blinded Reading) and the Semiquantitative (MPRI; Expert Evaluation) Gadobutrol Perfusion MRI Diagnosis Based on Myocardial Regions
Description: Rest and stress perfusion MR images were visually evaluated by 3 blinded readers. The MPRI was calculated by an independent MR expert. Analysis was performed for 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA): Visual and semiquantitative data were compared to each other per region. The number of regional assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial regions.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Regional Assessments) | 396 | 513 | 477 | 477
Percent regional assessments
  Disagreement | 56.3 | 55.2 | 49.1 | 58.3
  Agreement | 43.7 | 44.8 | 50.9 | 41.7

27. Secondary Outcome: Percentage Agreement Between the Visual (Blinded Reading) and Semiquantitative (MPRI; Expert Evaluation) Gadobutrol Perfusion MRI Diagnosis Based on Myocardial Segments
Description: Rest and stress perfusion MR images were visually evaluated by 3 blinded readers. The MPRI was calculated by an independent MR expert. Analysis was performed for 16 myocardial segments (defined according to the American Heart Association). Visual and semiquantitative data were compared to each other per segment. The number of segmental assessments was calculated by multiplication of the number of participants with the number of the blinded readers and the number of the myocardial segments.
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segmental Assessments) | 2112 | 2736 | 2544 | 2544
Percent segmental assessments
  Disagreement | 53.0 | 46.3 | 41.8 | 43.7
  Agreement | 47.0 | 53.7 | 58.2 | 56.3

28. Secondary Outcome: Signal Intensity (SIrel) Based on Segments
Description: The signal intensity (SIrel) is determined over time. SI (SIrel) is the upslope in myocardium divided by upslope of the ventricle, as assessed for normal and underperfused segments. SI(rel) = upslope myocard / upslope ventricle. MR segments were evaluated for signal intensity (SIrel) in order to assess if a difference between normal and diseased (i.e. ischemia/scar/mixed) segments could be demonstrated ("normal/diseased" was defined by central reading of SPECT).
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Mean (Standard Deviation); unit: Signal intensity
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Signal intensity
  Normal segment | 0.768 (2.0791) | 0.625 (0.3992) | 0.708 (0.8233) | 0.615 (0.2428)
  Disease segment | 0.732 (1.5511) | 0.603 (0.5428) | 0.813 (2.0755) | 0.584 (0.2424)

29. Secondary Outcome: Upslope Based on Segments
Description: "Upslope" is defined as the maximum slope of the signal intensity (SI) increase on the SI/time curve (determined by a linear fit) during 3 consecutive heart beats reported in "Units/sec". The upslope was evaluated for normal and for diseased (i.e. ischemia/scar/mixed) segments in order to assess a potential difference ("normal/diseased" was defined by central reading of SPECT).
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: PPS
Measure: Mean (Standard Deviation); unit: Units/sec
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Units/sec
  Normal segment | 11.44 (7.389) | 18.18 (9.850) | 27.49 (17.704) | 31.31 (24.339)
  Disease segment | 11.41 (6.730) | 17.90 (8.587) | 22.13 (13.997) | 26.93 (19.890)

30. Secondary Outcome: Time to Peak Based on Segments
Description: "Time to peak" is defined as the time in seconds from start to maximum signal intensity (SI max) on the SI curve and was evaluated for normal and for diseased (i.e. ischemia/scar/mixed) segments in order to assess a potential difference (normal/diseased was defined by central reading of SPECT).
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration up to 2 minutes
Population: PPS
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Seconds
  Normal segment | 12.43 (4.241) | 13.83 (4.407) | 13.87 (4.636) | 15.34 (4.403)
  Disease segment | 12.11 (3.796) | 13.67 (4.104) | 15.75 (4.982) | 16.34 (4.519)

31. Secondary Outcome: Percentage Agreement Between Presence/Absence of Delayed Enhancement in MRI (Blinded Reading) and Scar in SPECT (Central Reading) Based on Myocardial Regions
Description: Delayed enhancement (DE) -[accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions]- MR images acquired at different time points, were evaluated by 3 independent blinded readers for presence/absence of DE at 5 - 20 minutes post injection in 3 myocardial regions representing the 3 arterial territories of the heart. DE data were compared to the diagnosis "scar" derived from SPECT. The number of regional assessments is defined as the number of regions with diagnosis "scar" assessed by at least 1 blinded reader.
Time Frame: Delayed enhancement was measured at 5, 10, 15, and 20 minutes after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. Only participants with the finding "scar" in at least 1 segment in SPECT were included.
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 12 | 19 | 13 | 19
Number analyzed (Regional Assessments) | 48 | 72 | 42 | 96
Percent regional assessments
  region - 5 min DE | 0.0 | 1.4 | 14.3 | 36.5
  region - 10 min DE | 0.0 | 5.6 | 19.0 | 33.3
  region - 15 min DE | 0.0 | 2.8 | 19.0 | 38.5
  region - 20 min DE | 0.0 | 2.8 | 19.0 | 39.6

32. Secondary Outcome: Percentage Agreement Between Presence/Absence of Delayed Enhancement in MRI (Blinded Reading) and Scar in SPECT (Central Reading) Based on Myocardial Segments
Description: Delayed enhancement -[accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions]- MR images acquired at different time points were evaluated by 3 independent blinded readers regarding the presence/absence of DE at 5 - 20 minutes post injection in 16 myocardial segments (defined according to the American Heart Association). DE data were compared to the diagnosis "scar" derived from SPECT. The number of segmental assessments is defined as the number of segments with diagnosis "scar" assessed by at least 1 blinded reader.
Time Frame: Delayed enhancement was measured at 5, 10, 15, and 20 minutes after Gadobutrol bolus administration
Population: as for outcome 31
Measure: Number; unit: Percent segmental assessments
Units Other Than Participants: Segmental Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 12 | 19 | 13 | 19
Number analyzed (Segmental Assessments) | 129 | 147 | 111 | 195
Percent segmental assessments
  segment - 5 min DE | 0.0 | 0.7 | 18.9 | 31.3
  segment - 10 min DE | 0.0 | 2.7 | 20.7 | 28.7
  segment - 15 min DE | 0.0 | 1.4 | 20.7 | 35.4
  segment - 20 min DE | 0.0 | 1.4 | 20.7 | 36.4

33. Secondary Outcome: Percentage Agreement Between Presence/Absence of Delayed Enhancement in MRI (Clinical Evaluation) and Scar in SPECT (Central Reading) Based on Myocardial Regions
Description: Delayed enhancement (DE) -[accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions]- MR images acquired at different time points, were evaluated by the clinical investigator for presence/absence of DE at 5 - 20 minutes post injection in 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA). DE data were compared to the diagnosis "scar" derived from SPECT. The number of regional assessments is defined as the number of regions with diagnosis "scar" assessed by the investigator.
Time Frame: Delayed enhancement was measured at 5, 10, 15, and 20 minutes after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. Only participants with the finding "scar" in at least 1 region in SPECT were included.
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 12 | 19 | 13 | 19
Number analyzed (Regional Assessments) | 16 | 24 | 14 | 32
Percent regional assessments
  region - 5 min DE | 6.3 | 4.2 | 21.4 | 25.0
  region - 10 min DE | 6.3 | 4.2 | 28.6 | 37.5
  region - 15 min DE | 6.3 | 12.5 | 28.6 | 37.5
  region - 20 min DE | 6.3 | 4.2 | 21.4 | 37.5

34. Secondary Outcome: Percentage Agreement Between Presence/Absence of Delayed Enhancement in MRI (Clinical Evaluation) and Scar in SPECT (Central Reading) Based on Myocardial Segments
Description: Delayed enhancement (DE)-[accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions]- MR images acquired at different time points were evaluated by the respective investigator regarding the presence/absence of delayed enhancement at 5 - 20 minutes post injection in 16 myocardial segments (defined according to the American Heart Association). DE data were compared to the diagnosis "scar" derived from SPECT. The number of segmental assessments is defined as the number of segments with diagnosis "scar" assessed by the investigator.
Time Frame: Delayed enhancement was measured at 5, 10, 15, and 20 minutes after Gadobutrol bolus administration
Population: as for outcome 31
Measure: Number; unit: Percent segmental assessment
Units Other Than Participants: Segmental Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 12 | 19 | 13 | 19
Number analyzed (Segmental Assessment) | 43 | 49 | 37 | 65
Percent segmental assessment
  segment - 5 min DE | 4.7 | 2.0 | 21.6 | 23.1
  segment - 10 min DE | 7.0 | 2.0 | 24.3 | 30.8
  segment - 15 min DE | 9.3 | 6.1 | 18.9 | 32.3
  segment - 20 min DE | 2.3 | 2.0 | 18.9 | 30.8

35. Secondary Outcome: Assessment of the Overall Confidence in the Presence of Delayed Enhancement (DE) at 5 Minutes Post Injection (Blinded Reading)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions. Results are displayed on a per patient basis.
Time Frame: Delayed enhancement was measured at 5 minutes after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. The evaluation included only participants with delayed enhancement in at least 1 segment ( PPS) based on the assessment of at least one blinded reader.
Measure: Number; unit: Delayed enhancement assessments
Units Other Than Participants: Delayed enhancement assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 5 | 8 | 19 | 20
Number analyzed (Delayed enhancement assessments) | 5 | 14 | 40 | 49
Delayed enhancement assessments
  Poor | 5 | 12 | 11 | 8
  Satisfactory | 0 | 1 | 6 | 15
  good/excellent | 0 | 1 | 23 | 26

36. Secondary Outcome: Assessment of the Overall Confidence in the Presence of Delayed Enhancement (DE) at 5 Minutes Post Injection (Clinical Evaluation) (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 5 minutes after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. Evaluation includes only participants with delayed enhancement in at least 1 segment.
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 2 | 10 | 13 | 16
Participants
  Poor | 1 | 4 | 1 | 4
  Satisfactory | 0 | 4 | 4 | 2
  Good/excellent | 1 | 2 | 8 | 10

37. Secondary Outcome: Assessment of the Overall Confidence in the Presence of Delayed Enhancement (DE) at 10 Minutes Post Injection (Blinded Reading) (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions. Assessments of participants and/or segments by the individual blinded readers could differ. For the average reader, the results of the 3 individual readers are summarized
Time Frame: Delayed enhancement was measured at 10 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Delayed enhancement assessments
Units Other Than Participants: Delayed enhancement assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 3 | 10 | 19 | 23
Number analyzed (Delayed enhancement assessments) | 3 | 20 | 40 | 51
Delayed enhancement assessments
  Poor | 3 | 11 | 14 | 14
  Satisfactory | 0 | 5 | 3 | 12
  Good/excellent | 0 | 4 | 23 | 25

38. Secondary Outcome: Assessment of the Overall Confidence in the Presence of Delayed Enhancement (DE) at 10 Minutes Post Injection (Clinical Evaluation) (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 10 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 5 | 14 | 17 | 17
Participants
  Poor | 1 | 6 | 2 | 3
  Satisfactory | 2 | 3 | 3 | 2
  Good/excellent | 2 | 5 | 12 | 12

39. Secondary Outcome: Assessment of the Overall Confidence in the Presence of Delayed Enhancement (DE) at 15 Minutes Post Injection (Blinded Reading) (Only Participants With DE in at Least One Segment, PPS)
Description: as for outcome 37
Time Frame: Delayed enhancement was measured at 15 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Delayed enhancement assessments
Units Other Than Participants: Delayed enhancement assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 3 | 8 | 18 | 24
Number analyzed (Delayed enhancement assessments) | 3 | 15 | 44 | 56
Delayed enhancement assessments
  Poor | 3 | 8 | 15 | 17
  Satisfactory | 0 | 4 | 6 | 11
  Good/excellent | 0 | 3 | 23 | 28

40. Secondary Outcome: Assessment of the Overall Confidence in the Presence of Delayed Enhancement (DE) at 15 Minutes Post Injection (Clinical Evaluation) (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 15 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 5 | 12 | 17 | 17
Participants
  Poor | 2 | 5 | 2 | 4
  Satisfactory | 2 | 4 | 6 | 1
  Good/excellent | 1 | 3 | 9 | 12

41. Secondary Outcome: Assessment of the Overall Confidence in the Presence of Delayed Enhancement (DE) at 20 Minutes Post Injection (Blinded Reading) (Only Participants With DE in at Least One Segment, PPS)
Description: as for outcome 37
Time Frame: Delayed enhancement was measured at 20 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Delayed enhancement assessments
Units Other Than Participants: Delayed enhancement assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 4 | 11 | 20 | 25
Number analyzed (Delayed enhancement assessments) | 5 | 19 | 44 | 60
Delayed enhancement assessments
  Poor | 5 | 11 | 15 | 18
  Satisfactory | 0 | 4 | 10 | 17
  Good/excellent | 0 | 4 | 19 | 25

42. Secondary Outcome: Assessment of the Overall Confidence in the Presence of Delayed Enhancement (DE) at 20 Minutes Post Injection (Clinical Evaluation) (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 20 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 5 | 11 | 15 | 16
Participants
  Poor | 4 | 3 | 1 | 3
  Satisfactory | 1 | 5 | 5 | 0
  Good/excellent | 0 | 3 | 9 | 13

43. Secondary Outcome: Assessment of Contrast Quality of Delayed Enhancement (DE) at 5 Minutes Post Injection (Blinded Reading) (Only Participants With DE in at Least One Segment, PPS)
Description: as for outcome 37
Time Frame: Delayed enhancement was measured at 5 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Delayed enhancement assessments
Units Other Than Participants: Delayed enhancement assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 5 | 8 | 19 | 20
Number analyzed (Delayed enhancement assessments) | 5 | 14 | 40 | 49
Delayed enhancement assessments
  Poor | 5 | 11 | 13 | 8
  Satisfactory | 0 | 2 | 3 | 20
  Good/excellent | 0 | 1 | 24 | 21

44. Secondary Outcome: Assessment of Contrast Quality of Delayed Enhancement (DE) at 5 Minutes Post Injection (Clinical Evaluation) (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 5 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 2 | 10 | 13 | 16
Participants
  Poor | 2 | 3 | 3 | 4
  Satisfactory | 0 | 5 | 3 | 1
  Good/excellent | 0 | 2 | 7 | 11

45. Secondary Outcome: Assessment of Contrast Quality of Delayed Enhancement (DE) at 10 Minutes Post Injection (Blinded Reading) (Only Participants With DE in at Least One Segment, PPS)
Description: as for outcome 37
Time Frame: Delayed enhancement was measured at 10 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Delayed enhancement assessments
Units Other Than Participants: Delayed enhancement assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 4 | 10 | 19 | 23
Number analyzed (Delayed enhancement assessments) | 4 | 20 | 40 | 51
Delayed enhancement assessments
  Poor | 4 | 13 | 13 | 15
  Satisfactory | 0 | 5 | 5 | 15
  Good/excellent | 0 | 2 | 22 | 21

46. Secondary Outcome: Assessment of Contrast Quality of Delayed Enhancement (DE) at 10 Minutes Post Injection According to Clinical Evaluation (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 10 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 5 | 14 | 17 | 17
Participants
  Poor | 1 | 5 | 3 | 3
  Satisfactory | 1 | 5 | 2 | 2
  Good/excellent | 3 | 4 | 12 | 12

47. Secondary Outcome: Assessment of Contrast Quality of Delayed Enhancement (DE) at 15 Minutes Post Injection According to Blinded Reading (Only Participants With DE in at Least One Segment, PPS)
Description: as for outcome 37
Time Frame: Delayed enhancement was measured at 15 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Delayed enhancement assessments
Units Other Than Participants: Delayed enhancement assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 4 | 8 | 18 | 24
Number analyzed (Delayed enhancement assessments) | 4 | 15 | 44 | 56
Delayed enhancement assessments
  Poor | 4 | 11 | 13 | 15
  Satisfactory | 0 | 2 | 11 | 16
  Good/excellent | 0 | 2 | 20 | 25

48. Secondary Outcome: Assessment of Contrast Quality of Delayed Enhancement (DE) at 15 Minutes Post Injection According to Clinical Evaluation (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 15 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 5 | 12 | 17 | 17
Participants
  Poor | 3 | 4 | 3 | 4
  Satisfactory | 1 | 5 | 4 | 1
  Good/excellent | 1 | 3 | 10 | 12

49. Secondary Outcome: Assessment of Contrast Quality of Delayed Enhancement (DE) at 20 Minutes Post Injection According to Blinded Reading (Only Participants With DE in at Least One Segment, PPS)
Description: as for outcome 37
Time Frame: Delayed enhancement was measured at 20 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Delayed enhancement assessments
Units Other Than Participants: Delayed enhancement assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 4 | 11 | 20 | 25
Number analyzed (Delayed enhancement assessments) | 5 | 19 | 44 | 60
Delayed enhancement assessments
  Poor | 5 | 12 | 12 | 14
  Satisfactory | 0 | 4 | 18 | 25
  Good/excellent | 0 | 3 | 14 | 21

50. Secondary Outcome: Assessment of Contrast Quality of Delayed Enhancement (DE) at 20 Minutes Post Injection According to Clinical Evaluation (Only Participants With DE in at Least One Segment, PPS)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 20 minutes after Gadobutrol bolus administration
Population: as for outcome 36
Measure: Number; unit: Participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 5 | 11 | 15 | 16
Participants
  Poor | 4 | 2 | 2 | 3
  Satisfactory | 1 | 5 | 3 | 1
  Good/excellent | 0 | 4 | 10 | 12

51. Secondary Outcome: Percent Agreement Between Gadobutrol Perfusion MRI Diagnosis (Blinded Reading) and the Presence/Absence of Delayed Enhancement (DE) at the Time Point of Highest Agreement Between SPECT (Central Reading) and DE Based on Myocardial Regions
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions. Rest and stress perfusion MR and DE images were evaluated by 3 blinded readers for absence/presence of "scar" on perfusion MR and presence/absence of DE on MR for 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA).
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in PPS with assessment for this outcome measure. Evaluation included all participants in the per protocol population with an assessment for this outcome measure.
Measure: Number; unit: Percent regional assessments
Units Other Than Participants: Regional Assessments
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 0 | 37 | 25 | 26
Number analyzed (Regional Assessments) | 0 | 91 | 52 | 69
Percent regional assessments |  | 12.1 | 21.2 | 27.5

52. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI Diagnosis (Blinded Reading) and the Presence/Absence of Delayed Enhancement (DE) at the Time Point of Highest Agreement Between SPECT (Central Reading) and DE Based on Myocardial Segments
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions. Rest and stress perfusion MR and DE images were evaluated by 3 blinded readers for absence/presence of "scar" on perfusion MR and presence/absence of DE on MR for 16 myocardial segments (defined according to AHA).
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: as for outcome 51
Measure: Number; unit: Percent segmental assessment
Units Other Than Participants: Segmental Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 0 | 37 | 25 | 26
Number analyzed (Segmental Assessment) | 0 | 179 | 85 | 126
Percent segmental assessment |  | 7.3 | 27.1 | 23.8

53. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI Diagnosis (Clinical Evaluation) and the Presence/Absence of Delayed Enhancement (DE) at the Time Point of Highest Agreement Between SPECT (Central Reading) and DE Based on Myocardial Segments
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions. Rest and stress perfusion MR and DE images were evaluated by the clinical investigator for absence/presence of "scar" on perfusion MR and presence/absence of DE on MR for 16 myocardial segments (defined according to AHA).
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: as for outcome 51
Measure: Number; unit: Percent segmental assessment
Units Other Than Participants: Segmental Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 3 | 8 | 9 | 9
Number analyzed (Segmental Assessment) | 12 | 20 | 34 | 23
Percent segmental assessment | 41.7 | 75.0 | 82.4 | 100.0

54. Secondary Outcome: Percentage Agreement Between Gadobutrol Perfusion MRI Diagnosis (Clinical Evaluation) and Presence/Absence of Delayed Enhancement (DE) at the Time Point of Highest Agreement Between SPECT (Central Reading) and DE Based on Myocardial Regions
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions. Rest and stress perfusion MR and DE images were evaluated by the clinical investigator for absence/presence of "scar" on perfusion MR and presence/absence of DE on MR for 3 myocardial regions representing the 3 coronary territories/arteries (LAD, LCX, RCA).
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: as for outcome 51
Measure: Number; unit: Percent regional assessment
Units Other Than Participants: Regional Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 3 | 8 | 9 | 9
Number analyzed (Regional Assessment) | 5 | 11 | 16 | 14
Percent regional assessment | 20.0 | 72.7 | 87.5 | 92.9

55. Secondary Outcome: Percentage of Segments With Artifacts on Delayed Enhancement Images (Blinded Reading)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 5, 10, 15, and 20 minutes after Gadobutrol bolus administration
Population: PPS. Evaluation included all participants in the per protocol population with an assessment for this outcome measure
Measure: Number; unit: Percent segmental assessment
Units Other Than Participants: Segmental Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 57 | 53 | 53
Number analyzed (Segmental Assessment) | 2112 | 2736 | 2544 | 2544
Percent segmental assessment
  5 min DE | 23.9 | 22.3 | 26.7 | 26.2
  10 min DE | 25.3 | 19.4 | 18.2 | 22.6
  15 min DE | 20.9 | 18.0 | 20.7 | 24.7
  20 min DE | 19.2 | 16.4 | 18.7 | 21.8

56. Secondary Outcome: Percentage of Segments With Artifacts on Delayed Enhancement Images (Clinical Evaluation)
Description: Delayed enhancement: accumulation of Gadobutrol in infarcted tissue and visualized as Gadobutrol enhanced regions.
Time Frame: Delayed enhancement was measured at 5, 10, 15, and 20 minutes after Gadobutrol bolus administration
Population: as for outcome 51
Measure: Number; unit: Percent segmental assessment
Units Other Than Participants: Segmental Assessment
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 44 | 55 | 53 | 53
Number analyzed (Segmental Assessment) | 704 | 880 | 848 | 848
Percent segmental assessment
  5 min DE | 26.8 | 24.9 | 21.3 | 11.7
  10 min DE | 23.3 | 21.3 | 10.6 | 13.8
  15 min DE | 23.7 | 19.4 | 13.7 | 11.9
  20 min DE | 24.9 | 22.8 | 13.4 | 14.2

57. Secondary Outcome: Percentage of Participants With Deviation of MRI Procedure (Clinical Evaluation)
Time Frame: Immediately within approximately 5 seconds after Gadobutrol bolus administration
Population: All participants in FAS with assessment for this outcome measure. Evaluation included all participants in the full analysis population with an assessment for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Number analyzed (Participants) | 52 | 60 | 56 | 54
Percentage of participants
  No | 86.5 | 76.7 | 76.8 | 85.2
  Yes | 13.5 | 23.3 | 23.2 | 14.8

ADVERSE EVENTS:
Arm/Group | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875)
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/60 | 0/58 | 0/54
Other Adverse Events (participants affected / at risk) | 3/54 | 1/60 | 4/58 | 5/54
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol 0.01 mmol/kg BW (Gadavist, BAY86-4875) (N=54) | Gadobutrol 0.025 mmol/kg BW (Gadavist, BAY86-4875) (N=60) | Gadobutrol 0.05 mmol/kg BW (Gadavist, BAY86-4875) (N=58) | Gadobutrol 0.1 mmol/kg BW (Gadavist, BAY86-4875) (N=54)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study designed for perfusion imaging, not optimized for delayed enhancement. Routine SPECT selected as standard of reference (SoR) despite known quality limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less